CLINICAL TRIAL: NCT00162773
Title: Effect of Anti-IgE in Non-Allergic Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-10-25-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): water injection
  Interventions: Other: Placebo
- Omalizumab (Experimental): Other Names:
  Xolair 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
  Other Names: Xolair
  Arms: Omalizumab
Other: Placebo — 150-375 milligrams depending on body weight and serum IgE.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if omalizumab is effective in treating non-allergic asthma. The US Food and Drug Administration has approved the use of omalizumab to treat moderate to severe allergic asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease of the lower airways. The inflammatory process is associated with changes in airway hyperresponsiveness (irritability), and airflow limitations caused by bronchoconstriction, edema, and mucous plugging. Mast cells, basophils, eosinophils, activated T-lymphocytes, macrophages, neutrophils, and airway epithelial cells all play a role in this inflammatory process by releasing mediators directly responsible for local inflammation and by releasing mediators that encourage a further influx of inflammatory cells (Expert Panel Report 2, 1997). These cells and their products eventually produce a state of chronic allergic inflammation leading to increased vascular leakage, mucous secretion, smooth muscle hyperresponsiveness, and nerve activation. Clinically, this process is characterized by intermittent shortness of breath, wheezing, coughing, and chest tightness.

Although most asthmatics are atopic (allergic), non-atopic asthmatics exist and can develop equally severe disease. Non-allergic asthmatics have a trend towards higher than normal levels of the allergic antibody (IgE) though obviously they lack skin test specificity. When examining skin test reactivity and serum IgE as independent variables for asthma risk, there was a stronger association with serum IgE elevation than skin test reactivity. In fact, serum IgE tended to be high in asthmatics regardless of skin test reactivity.

Omalizumab (Xolair®) is a recombinant humanized monoclonal antibody that binds specifically to the (FceRI) binding site on human IgE. The binding of omalizumab inhibits the ability of IgE to bind to basophils or mast cells.

Omalizumab recently received FDA approval for the treatment of moderate to severe persistent allergic asthma in pediatric (12 years of age and above) and adult patients. The addition of omalizumab to standard asthma therapies has been found to reduce asthma exacerbations and decrease both inhaled corticosteroid dose and rescue medication use. (Busse, 2001). In a phase III double blinded placebo controlled trial involving 525 severe allergic asthmatics, omalizumab treated patients had fewer exacerbations during both a steroid stable phase and steroid reduction phase than did placebo controls (Busse, 2001). The median reduction in steroid dose during reduction phase was 75% and 50% in the omalizumab and placebo groups respectively. In a similarly designed steroid reduction study involving 6 to 12 year-old moderate to severe allergic asthmatics, steroid reduction was possible in 100% of treated patient verses 66.7% of placebo treated patients (Milgrom, 2001). Other steroid reduction studies have had similar results (Buhl 2002, Soler 2001). Omalizumab has also been shown to improve quality of life in allergic asthmatics as measured by the Asthma Quality of Life Questionnaire (AQLQ). In adults, AQLQ demonstrated greater improvement at 16, 28 and 52 weeks in omalizumab treated patients than in placebo treated (Finn 2003). Similarly in pediatric populations, AQLQ improvement reached statistical significance in omalizumab treated patients (Lemanske 2002).

Omalizumab has shown itself to be a promising new therapy for the treatment of moderate to severe allergic asthma. It is currently not indicated for patients with non-allergic asthma. The objective of this study will be to define the effects of omalizumab on cell surface FceRI expression and serum IgE of non-allergic asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-breastfeeding females 18 through 80 years of age
* Clinically acceptable ECG
* Diagnosis of moderate to severe persistent asthma
* History or presence of episodic symptoms of airflow obstruction (wheeze, chest tightness, cough, shortness of breath)
* Airflow obstruction is at least partially reversible
* FEV1 in the context of this study is <80%of predicted values at visit 1 with no short-acting ß agonist use within 6 hours of spirometry
* Improvement of at least 12% of predicted FEV1 value and at least 200 ml within 15 to 30 minutes of inhaling nebulized albuterol (up to 5mg) or 2-4 puffs of albuterol (90 mcg/actuation) demonstrated at study entry or documented in the last year.
* Subjects must be able to demonstrate proper technique for use of the MiniWright peak flow meter
* Subjects must have a negative skin test to the 5 common perennial aeroallergens (D. farinae, D. pteronyssinus, cat, dog, and cockroach) at prick puncture with an adequate histamine control.
* Subjects must have negative RAST to the same 5 common perennial aeroallergens .
* Serum total IgE must be 30-700 IU/ml.
* Normal EKG at baseline
* Females must be: Surgically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation), OR postmenopausal (at least 1 year since last menses), OR using one of the following medically acceptable forms of birth control throughout the duration of the study:

  * Systemic contraceptives
  * Diaphragm with intravaginal spermicide
  * Cervical cap
  * Intrauterine device
  * Condom with intravaginal spermicide
* Females in certain categories (not sexually active, vasectomized partner) will be admitted at the discretion of the investigator on a case-by-case basis. Accepted cases will be documented on the Female Enrollment Form and kept with the informed consent document.
* Females, excluding those more than 1 year postmenopausal or who are surgically sterile, must have a negative urine pregnancy test at Visit 1 and other visits specified in this protocol. If a subject becomes pregnant during the study participation, they will be discharged from the study and followed until termination of the pregnancy or delivery is complete.

Exclusion Criteria:

* Respiratory tract infection within 14 days prior to Visit 1
* Chronic bronchitis, COPD, emphysema and other chronic lung diseases
* Receiving immunotherapy other than maintenance therapy
* Current smokers
* Current use of Xolair®
* Recent history of drug or alcohol abuse (within 3 years prior to Visit 1)
* Pregnant or likely to become pregnant during the study
* Breast-feeding
* History of hypersensitivity to albuterol, or Xolair, or to drugs with similar chemical structures
* Treatment with any investigational drug in the last 30 days before enrollment into the study (Visit 1)
* Clinically relevant cardiovascular, hepatic, neurologic, psychiatric, endocrine, or other major systemic disease making the protocol or interpretation of the study results difficult
* Site staff members or their immediate families are not eligible to enroll

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Creticos, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The arms/groups were combined for the study due to the study's early termination and the PI's departure from the institution. Data obtained were from the IRB and are therefore not separated by arm. This is all that is available.
Groups:
- All Participants: water injection/Placebo: 150-375 milligrams depending on body weight and serum IgE.
  OR
  Other Names:
  Xolair/Omalizumab 150-375 milligrams administered by subcutaneous injection every 2-4 weeks
Period: Overall Study
Arm/Group | All Participants
Started | 29
Completed | 7
Not Completed | 22
Not completed — P.I, Left institution. Study terminated | 22

BASELINE CHARACTERISTICS:
Groups:
- All Participants: water injection/Placebo: 150-375 milligrams depending on body weight and serum IgE.
  OR
  Other Names:
  Xolair/Omalizumab 150-375 milligrams administered by subcutaneous injection every 2-4 weeks omalizumab: 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Customized [Count of Participants; unit: Participants]
  >=18 and <=80 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Changes in Free Serum IgE Levels From Baseline
Time Frame: baseline to 2 weeks
Population: Data, if any, are not available as this study has been terminated as the PI has left the institution. The arms/groups were combined for the study due to the study's early termination and the PI's departure from the institution. Data obtained were from the IRB and are therefore not separated by arm. This is all that is available.
Groups:
- All Participants: water injection
  Placebo: 150-375 milligrams depending on body weight and serum IgE.
  OR
  Other Names:
  Xolair 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
  omalizumab: 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The arms/groups were combined for the study due to the study's early termination and the PI's departure from the institution. Data obtained were from the IRB and are therefore not separated by arm. This is all that is available.
Groups:
- All Participants: water injection/Placebo: 150-375 milligrams depending on body weight and serum IgE.
  OR
  Xolair/Omalizumab 150-375 milligrams administered by subcutaneous injection every 2-4 weeks depending on body weight and serum IgE.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=29)
Boil/Abscess/Cellulitis (Infections and infestations) | 1 (1) — One participant developed a skin and soft tissue infection at the injection site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes